CLINICAL TRIAL: NCT02413593
Title: A Phase 2 Open- Label Study to Evaluate The Safety and Efficacy of Ledipasvir/Sofosbuvir (LDV/SOF) Fixed Dose Combination Tablet With Ribavirin for 12 Weeks in Treatment-naïve Patients With Chronic HCV Genotype 3 Infection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir (LDV/SOF) Fixed Dose Combination Tablet With Ribavirin for 12 Weeks in Treatment-naive Adults With Chronic HCV Genotype 3 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1701
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2016-12

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV genotype 3 (GT-3); HCV; Sustained Virologic Response; Direct Acting Antiviral; GS-7977; GS-5885; Ribavirin; Sofosbuvir; Ledipasvir; Hepatitis C; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDV/SOF+RBV (Experimental): LDV/SOF FDC plus RBV for 12 weeks
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study will evaluate the antiviral efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed dose combination (FDC) plus ribavirin (RBV) in treatment-naive adults with chronic genotype 3 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic genotype 3 HCV infection
* HCV treatment-naive
* HCV RNA > 10,000 IU/mL at screening
* Absence of cirrhosis or compensated cirrhosis
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Key Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Coinfection with HIV or hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with the individual's treatment, assessment, or compliance with the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (10):
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brampton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Vaughan, Ontario
  - Montreal, Quebec
  - Québec

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Feld JJ, Ramji A, Shafran S, Willems B, Marotta P, Huchet E, et al. Ledipasvir/Sofosbuvir with ribavirin for 12 Weeks is effective and safe in treatment-naïve genotype 3 HCV-infected patients in Canada [Abstract SAT-183]. Presented at: The 51st Annual Congress of the European Association for the Study of Liver: The International Liver Congress (EASL); 2016 April 13-17; Barcelona, Spain.
- [Derived] Feld JJ, Ramji A, Shafran SD, Willems B, Marotta P, Huchet E, Vachon ML, Svarovskaia ES, Huang KC, Hyland RH, Yun C, Massetto B, Brainard DM, McHutchison JG, Tam E, Bailey R, Cooper C, Yoshida EM, Greenbloom S, Elkhashab M, Borgia S, Swain MG. Ledipasvir-Sofosbuvir Plus Ribavirin in Treatment-Naive Patients With Hepatitis C Virus Genotype 3 Infection: An Open-Label Study. Clin Infect Dis. 2017 Jul 1;65(1):13-19. doi: 10.1093/cid/cix289. PMID 28535298

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Canada. The first participant was screened on 15 April 2015. The last study visit occurred on 08 January 2016.
Pre-assignment Details: 127 participants were screened.
Groups:
- LDV/SOF+RBV: Ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks
Period: Overall Study
Arm/Group | LDV/SOF+RBV
Started | 111
Completed | 107
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study drug.
Groups:
- LDV/SOF+RBV: LDV/SOF (90/400 mg) FDC tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
Arm/Group | LDV/SOF+RBV
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 111
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 78
  More than one race | 1
  Unknown or Not Reported | 0
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 3 (no confirmed subtype) | 3
  Genotype 3a | 105
  Genotype 3b | 3
Cirrhosis Status [Count of Participants; unit: Participants]
  Absent | 70
  Present | 39
  Missing | 2
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 40
    CT | 56
    TT | 13
    Missing | 2
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.66)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 35
  ≥ 800,000 IU/mL | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF+RBV
Number analyzed (Participants) | 111
percentage of participants | 89.2 [81.9 to 94.3]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV
Number analyzed (Participants) | 111
percentage of participants | 0.9

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF+RBV
Number analyzed (Participants) | 111
percentage of participants | 91.9 [85.2 to 96.2]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 1, 2, 4, 8 and 12
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF+RBV
Number analyzed (Participants) | 111
percentage of participants
  Week 1 | 20.7 [13.6 to 29.5]
  Week 2 | 64.9 [55.2 to 73.7]
  Week 4 | 97.3 [92.3 to 99.4]
  Week 8 | 100.0 [96.7 to 100.0]
  Week 12: number analyzed (Participants) | 110
  Week 12 | 99.1 [95.0 to 100.0]

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 8, and 12
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF+RBV
Number analyzed (Participants) | 111
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 110
  Change at Week 1 | -4.33 (0.572)
  Change at Week 2 | -4.85 (0.659)
  Change at Week 4 | -5.05 (0.664)
  Change at Week 8 | -5.06 (0.664)
  Change at Week 12: number analyzed (Participants) | 109
  Change at Week 12 | -5.06 (0.669)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF+RBV
Number analyzed (Participants) | 111
percentage of participants | 7.2

ADVERSE EVENTS:
Time Frame: Baseline to 30 days after last dose of study drug (up to 12 weeks plus 30 days)
Description: Safety Analysis Set
Arm/Group | LDV/SOF+RBV
Serious Adverse Events (participants affected / at risk) | 4/111
Other Adverse Events (participants affected / at risk) | 89/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF+RBV (N=111)
Hyponatraemia (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Homicidal ideation (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF+RBV (N=111)
Abdominal pain (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 57
Nasopharyngitis (Infections and infestations) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 40
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 19
Irritability (Psychiatric disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years